CLINICAL TRIAL: NCT06082102
Title: A Randomized, Controlled, Open-label, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of Orelabrutinib Plus Rituximab Versus Lenalidomide Plus Rituximab in Relapsed/Refractory Marginal Zone Lymphoma
Brief Title: Efficacy and Safety of Orelabrutinib Combined With Rituximab Versus Lenalidomide Combined With Rituximab in Patients With Relapsed/Refractory Marginal Zone Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00123
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — orelabrutinib; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orelabrutinib (Experimental)
  Interventions: Drug: Orelabrutinib; Drug: Rituximab
- Comparator (Active Comparator)
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib Tablets
  Arms: Orelabrutinib
Drug: Rituximab — Rituximab Injection
  Arms: Orelabrutinib
Drug: Lenalidomide — Lenalidomide Capsules
  Arms: Comparator
Drug: Rituximab — Rituximab Injection
  Arms: Comparator

SUMMARY:
Efficacy and Safety of Orelabrutinib Combined with Rituximab versus Lenalidomide Combined with Rituximab in Patients with Relapsed/Refractory Marginal Zone Lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years , either sex.
2. Histopathologically confirmed B-cell non-Hodgkin lymphoma MZL (splenic, nodal, or extra-nodal).
3. Prior systemic therapy including at least one anti-CD20 monoclonal antibody-containing regimen is required, with the following specifications:

   For combination therapies: Minimum of 2 completed treatment cycles For anti-CD20 monotherapy: Minimum of 4 administered doses Progression during treatment waives cycle/dose requirements
4. Relapsed or refractory disease.
5. At least 1 measurable lesion confirmed through enhanced computed tomography (CT) or enhanced magnetic resonance imaging (MRI).
6. ECOG performance status (PS) score of 0-2.

Exclusion Criteria:

1. Administration of the specified anti-tumor therapies within 2 weeks prior to the first dose of the study treatment.
2. Administration of any other investigational product within 4 weeks prior to the first dose of the study treatment, or concurrent participation in another clinical trial.(Excluding patients who have discontinued treatment and are in long-term follow-up).
3. Prior treatment with any types of BTK inhibitor.
4. Patients refractory to lenalidomide plus rituximab (R2 regimen). Refractoriness is defined as either: Failure to achieve at least partial response (PR) after completing an adequate R2 treatment course (≥2 cycles at standard doses), OR Disease progression during R2 therapy or within 6 months after the last dose.
5. Central nervous system (CNS) lymphoma, and lymphoma with CNS or meningeal involvements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2030-02-25 (Estimated)

PRIMARY OUTCOMES:
IRC-assessed PFS | Through study completion, an average of 5 year.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Auhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial Peoples Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The first Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital Of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University（Xibei Hospital）, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang